CLINICAL TRIAL: NCT01225029
Title: A Randomized Controlled Trial of Fluid Management in Transient Tachypnea of the Newborn
Brief Title: Fluid Management in Transient Tachypnea of the Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 07-1069
Record Dates: First submitted 2010-10-18; First posted 2010-10-20 (Estimated); Results first posted 2013-11-28 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-09

CONDITIONS: Transient Tachypnea of the Newborn
Keywords: premature birth; late preterm birth; respiratory distress of the newborn; Transient tachypnea of the newborn
MeSH Terms: conditions — Transient Tachypnea of the Newborn; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Fluids (No Intervention): Term neonates receive total fluids of 60 mL/kg/day on day of life (DOL) 1. Preterm neonates receive total fluids of 80 mL/kg/day on DOL 1. Each group receives an extra 20 mL/kg/day daily until total fluids of 150 mL/kg/day are achieved.
- Restricted Fluids (Experimental): Term neonates receive total fluids of 40 mL/kg/day on day of life (DOL) 1. Preterm neonates receive total fluids of 60 mL/kg/day on DOL 1. Each group receives an extra 20 mL/kg/day daily until total fluids of 150 mL/kg/day are achieved
  Interventions: Other: Amount of total fluids

INTERVENTIONS:
Other: Amount of total fluids — Term neonates receive either total fluids of 60 mL/kg/day (standard) or 40 mL/kg/day (restricted) on day of life (DOL) 1. Preterm neonates receive total fluids of 80 mL/kg/day (standard) or 60 mL/kg/day (restricted) on DOL 1. Each group receives an extra 20 mL/kg/day daily until total fluids of 150 mL/kg/day are achieved.
  Arms: Restricted Fluids

SUMMARY:
Transient tachypnea of the newborn (TTN) is a diagnosis given to infants born between 34 and 42 weeks gestation who develop difficulty breathing during the first days of life when no specific cause of the breathing difficulty can be identified. Little is known about why some babies develop TTN, and there have not been many formal studies of the best way to take care of babies with this disease. Babies with TTN get better on their own within three to five days after birth, but may require extra oxygen to breath well.

Most physicians believe that the symptoms of TTN are related to poor clearance of fluid from the newborn's lungs. Babies with TTN have extra fluid visible on chest x-ray. Diuretics, medicines that can help clear extra lung fluid in adults and in babies with extra lung fluid for other reasons, do not to help babies with TTN. Babies with TTN need intravenous fluids to be healthy because they breathe too fast to be able to eat. Breastfed babies only get a very small amount of fluid in the first few days of life, as it normally takes several days for a new mother to begin producing breastmilk. No one has yet examined whether giving babies with TTN an amount of fluid similar to the small amount they would receive if they could breastfeed would help them recover from TTN faster.

In this study, the investigators compare whether giving newborns "standard" intravenous fluid or amounts of intravenous fluid more close to what a breastfed baby would receive speeds recovery in newborns with TTN.

DETAILED DESCRIPTION:
1. Project Abstract Transient tachypnea of the newborn (TTN) is a self-limited respiratory distress syndrome of term and late pre-term neonates.1 Respiratory distress attributed to TTN requires management of otherwise healthy infants in an intensive care setting, thus increasing cost, and often length, of hospitalization as well as decreasing opportunity for parent-child bonding in the first days of life. Although hundreds of thousands of children are treated for TTN every year (over 250 in the Mount Sinai NICU in 2005 alone), little data underlie standard of care medical management. We are conducting a prospective study of neonates diagnosed with TTN to determine if changes in fluid management affects course of disease.
2. Specific Aims To determine whether fluid restriction in the first 72 hours of life speeds resolution of respiratory distress in neonates diagnosed with TTN.
3. Concise statement of Significance/Background Transient tachypnea of the newborn (TTN) is a self-limited respiratory distress syndrome of term and late pre-term neonates.1 Newborns with TTN develop clinical signs of respiratory distress within the first hours after birth, in the absence of other pathology such as surfactant deficiency, infection, meconium aspiration, or anatomic cardiac or pulmonary anomaly. Signs of TTN include tachypnea (respiratory rate consistently > 60), subcostal, intercostals, and suprasternal retractions, nasal flaring, grunting, and hypoxia correctable with low FiO2 supplemental oxygen (< 0.40) via conventional nasal cannula or continuous positive airway pressure (CPAP). The condition usually resolves with supportive care within 72 hours without significant long-term adverse sequelae. Transient tachypnea of the newborn is associated with transient pulmonary edema diagnosed by typical chest x-ray findings.

   The traditional explanation for postnatal pulmonary edema is poor clearance of fluid from the fetal lungs in the perinatal period. Retained fluid leads to bronchioalveolar collapse with variable areas of hyperinflation and air trapping in the neonatal lung. The newborn compensates for this ventilation/perfusion mismatch with tachypnea and increased work of breathing, but often cannot completely compensate, becoming hypoxic through the period of fluid reabsorption.

   This pathophysiologic argument has been supported by the findings that brief or absent labor and short or absent time in the birth canal have been associated with TTN.2, 3 It has long been hypothesized that mechanical forces of labor and delivery work to "squeeze" edema away from air-exchange surfaces of the lung into the lymphatics. More recently, studies have demonstrated that immaturity of sodium ion channel transporters in the lung epithelium may play a more significant role in the failure of pulmonary fluid reabsorption than mechanical forces.4, 5 Data from animal models show that absent labor, such as found in scheduled Cesarean sections, may lead to delivery before the normal hormonally-mediated upregulation or activation of these sodium transporters occurs and thus may explain the increased likelihood of developing TTN seen in this patient cohort.

   Conditions that increase central venous pressure or decrease thoracic duct clearance have also been associated with TTN.6 Additionally, maternal diagnosis of asthma7 or gestational diabetes8 and male gender of the newborn9 have been associated with TTN, although the mechanism of these associations is incompletely understood. Although TTN is an exceedingly common cause of newborn morbidity, it is relatively understudied. Due to the low mortality of TTN there has been little interest in investigating either the range of pathologies underlying the clinical presentation of TTN or the evidence base behind the standard of care treatments of TTN. The high incidence of TTN and the significant increase in hospital care acuity and length of stay to otherwise healthy infants diagnosed with TTN, however, indicates a need for study.10 As the rate of Cesarean section and late pre-term delivery,11 as well as maternal morbidities such as asthma12 and gestational diabetes,13 rise it is particularly important to minimize the morbidity and cost of TTN. A better understanding of the pathogenesis of TTN and a thorough evaluation of current treatment strategies and their relationship to timely patient discharge is sorely needed.
4. Concise statement of Preliminary Data (if available) No evidence base underlies current fluid management of neonates with TTN. Data exists demonstrating the inefficacy of loop diuretics as treatment for pulmonary fluid overload in newborns with TTN,14 but no systematic evaluation of intravenous fluid management exists. Exclusively breastfed babies typically have minimal fluid intake during the first four days of life as lactogenesis II (initial postpartum milk production) proceeds. Enteral intake by term infants begins at less than 100mL in the first day (equivalent to 40mL/kg for a 2.5kg neonate; this represents a term newborn at the 5th percentile or a 34 week gestational age newborn at the 70th percentile for weight) and increase gradually until milk production reaches sustenance levels, usually around the fourth day of life.15 Regardless of gestational age, all neonates lose water weight during the first week of life during physiologic diuresis of extracellular fluid accumulated throughout gestation.16 Current management of both preterm and term neonates includes an effort to facilitate this physiologic diuresis by gradually increasing amounts of IV fluids until maintenance levels are reached between the third and fifth day of life. 17, 18
5. Research Design and Methods In this study, we will conduct a prospective study of 68 neonates born between 34 and 42 weeks gestation diagnosed with TTN and managed in the Mount Sinai Neonatal Intensive Care Unit (NICU). The study period will include the first three days (72 hours) of life. On admission to the NICU, parents will be consented for their child's inclusion in the study. If consent is given, the child will be randomized to "standard fluids" or "physiologic fluids" groups. "Standard fluids" refer to current standard clinical practice of IV fluid administration, not based on experimental evidence. "Physiologic fluids" refers to IV fluid amounts more similar to fluid volumes typically ingested during initiation of breastfeeding. Term infants assigned to the "standard fluids" group will be started on 60 mL/kg/day of glucose-containing intravenous fluids as is standard practice. Term infants assigned to the "physiologic fluids" group will be started on 40 mL/kg/day glucose-containing intravenous fluids. Late preterm infants (gestational age between 34 and 37 weeks) assigned to the "standard fluids" group will be started on 80 mL/kg/day of glucose-containing intravenous fluids as is standard practice. Late preterm infants (gestational age between 34 and 37 weeks) assigned to the "physiologic fluids" group will be started on 60 mL/kg/day glucose-containing intravenous fluids. For all groups, intravenous fluid rate will be increased by 20 mL/kg/day daily, as is current standard practice. Consistent with current standard management for newborns with respiratory distress, no infant will be allowed to take oral nutrition until respiratory distress abates. Newborns will be carefully monitored, and infants in the "physiologic fluid" group will be removed from the study and total daily fluids will be increased if they show signs of dehydration. Primary outcomes will be duration of respiratory distress, defined as respiratory rate consistently greater than 50 breaths/minute and oxygen saturation on room air consistently less than 95%. Secondary outcomes will be length of time to first oral feed and time to discharge from the intensive care unit.

This research poses a minor increase over minimal risk for subjects enrolled in the intervention group. The anticipated risks include mild dehydration and/or hypoglycemia of neonates in the "physiologic fluid" intervention group. This risk is minor as all newborns in the NICU have urine output recorded every three hours, point-of-care glucose monitoring on admission and at least once every twelve hours thereafter, and serum electrolytes checked between 12 and 24 hours of life. If neonatal dehydration is noted as defined by urine output < 2mL/kg/hour over a twelve hour period, serum sodium < 130 mEq/L or > 150 mEq/L, weight loss of more than 10% of birth weight, or blood glucose by point-of-care testing of < 40 mg/dL, the child will be removed from the study and appropriate fluid resuscitation will be initiated. These guidelines for removal from the study are the same as or more conservative than criteria used for rehydration in clinical care, so long-term adverse sequelae of this level of brief mild dehydration or hypoglycemia are not expected.

ELIGIBILITY:
Inclusion Criteria:

1. Gestational age at birth 34 and 42 weeks of gestation
2. Admission to the Mount Sinai NICU during the first 24 hours of life
3. Diagnosis during the first 24 hours of life of transient tachypnea of the newborn

Exclusion criteria:

1. Gestational age at birth less than 34 weeks or greater than 42 weeks at birth
2. No diagnosis of TTN made in the first 24 hours of life
3. Additional infant diagnosis of major cardiac disease
4. Additional infant diagnosis of major pulmonary disease other than TTN
5. Additional infant diagnosis of meconium aspiration syndrome
6. Additional infant diagnosis of major congenital anomaly with potential to affect respiratory status in the neonatal period
7. Additional infant diagnosis of infectious disease process potentially affecting respiratory status in the neonatal period
8. Observation of thick meconium in the amniotic fluid at delivery.
9. Maternal diagnosis of chorioamnionitis or other infection of the uterus or fallopian tubes pre- or peri-partum.

Criteria for removal from the study:

(a) Additional infant diagnosis of major cardiac, pulmonary, or other disease process potentially affecting respiratory status in the neonatal period (i.e., infection, meconium aspiration, pneumothorax, congenital anomaly) present during the study period. (b) Positive test of infection (e.g. blood, CSF, or urine culture; viral DFA; microscopy) drawn from infant at any point during the study period. (c) Maternal diagnosis of chorioamnionitis or other infection of the uterus or fallopian tubes at any point during hospital stay. (d) Objective clinical signs of dehydration: (i) Newborn urine output less than 2 mL/kg/hr over a twelve hour period at any point during the study period. (ii) Newborn serum sodium less than 130 mEq/L or greater than 150 mEq/L at any point during the study period. (iii) Newborn weight loss >10% of birth weight at any point during the study period.

(e) Newborn blood glucose by point-of-care testing of less than 40 mg/dL at any point during the study period. (f) Administration of exogenous surfactant at any point during the study period.

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2008-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annemarie Stroustrup, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Avery ME, Gatewood OB, Brumley G. Transient tachypnea of newborn. Possible delayed resorption of fluid at birth. Am J Dis Child. 1966 Apr;111(4):380-5. doi: 10.1001/archpedi.1966.02090070078010. No abstract available. PMID 5906048
- [Background] Zanardo V, Simbi AK, Franzoi M, Solda G, Salvadori A, Trevisanuto D. Neonatal respiratory morbidity risk and mode of delivery at term: influence of timing of elective caesarean delivery. Acta Paediatr. 2004 May;93(5):643-7. doi: 10.1111/j.1651-2227.2004.tb02990.x. PMID 15174788
- [Background] Riskin A, Abend-Weinger M, Riskin-Mashiah S, Kugelman A, Bader D. Cesarean section, gestational age, and transient tachypnea of the newborn: timing is the key. Am J Perinatol. 2005 Oct;22(7):377-82. doi: 10.1055/s-2005-872594. PMID 16215925
- [Background] Jain L, Eaton DC. Physiology of fetal lung fluid clearance and the effect of labor. Semin Perinatol. 2006 Feb;30(1):34-43. doi: 10.1053/j.semperi.2006.01.006. PMID 16549212
- [Background] Jain L, Dudell GG. Respiratory transition in infants delivered by cesarean section. Semin Perinatol. 2006 Oct;30(5):296-304. doi: 10.1053/j.semperi.2006.07.011. PMID 17011402
- [Background] Demissie K, Marcella SW, Breckenridge MB, Rhoads GG. Maternal asthma and transient tachypnea of the newborn. Pediatrics. 1998 Jul;102(1 Pt 1):84-90. doi: 10.1542/peds.102.1.84. PMID 9651418
- [Background] Persson B, Hanson U. Neonatal morbidities in gestational diabetes mellitus. Diabetes Care. 1998 Aug;21 Suppl 2:B79-84. PMID 9704232
- [Background] Tutdibi E, Hospes B, Landmann E, Gortner L, Satar M, Yurdakok M, Dellagrammaticas H, Ors R, Ilikkan B, Ovali F, Sarman G, Kumral A, Arslanoglu S, Koc H, Yildiran A. Transient tachypnea of the newborn (TTN): a role for polymorphisms of surfactant protein B (SP-B) encoding gene? Klin Padiatr. 2003 Sep-Oct;215(5):248-52. doi: 10.1055/s-2003-42670. PMID 14520584
- [Background] Adams JM, Moreno J, Reynolds K, Campbell DW IV, Smith EO, Weisman LE. Resource utilization among neonatologists in a university children's hospital. Pediatrics. 1997 Jun;99(6):E2. doi: 10.1542/peds.99.6.e2. PMID 9164798
- [Background] Lewis V, Whitelaw A. Furosemide for transient tachypnea of the newborn. Cochrane Database Syst Rev. 2002;(1):CD003064. doi: 10.1002/14651858.CD003064. PMID 11869651
- [Background] Neville MC, Morton J. Physiology and endocrine changes underlying human lactogenesis II. J Nutr. 2001 Nov;131(11):3005S-8S. doi: 10.1093/jn/131.11.3005S. PMID 11694636
- [Derived] Stroustrup A, Trasande L, Holzman IR. Randomized controlled trial of restrictive fluid management in transient tachypnea of the newborn. J Pediatr. 2012 Jan;160(1):38-43.e1. doi: 10.1016/j.jpeds.2011.06.027. Epub 2011 Aug 11. PMID 21839467

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at our urban tertiary care center from August 1, 2008 through September 2, 2010. Patients were withdrawn from the study protocol if any respiratory diagnosis other than TTN was made.
Pre-assignment Details: 73 patients met enrollment criteria, and the parents of 67 eligible neonates agreed to participate. 34 were assigned to standard-of-care fluid management and 33 were assigned to the restricted fluid protocol. 2 patients from the standard fluid group and 1 patient from the restricted fluid group were withdrawn for a non-TTN respiratory diagnosis.
Groups:
- Standard Fluids: Term neonates receive total fluids of 60 mL/kg/day on day of life (DOL) 1. Each group receives an extra 20 mL/kg/day daily until total fluids of 150 mL/kg/day are achieved.
- Restricted Fluids: Preterm neonates receive total fluids of 60 mL/kg/day on DOL 1. Each group receives an extra 20 mL/kg/day daily until total fluids of 150 mL/kg/day are achieved
Period: Overall Study
Arm/Group | Standard Fluids | Restricted Fluids
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Fluids | Restricted Fluids | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Customized [Mean (Standard Deviation); unit: weeks] | 35.8 (1.6) | 36.4 (1.5) | 36.1 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 17 | 16 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 21 | 20 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Duration of Respiratory Support
Time Frame: every hour until patient stable without respiratory support, an average of approximately 55 hours and a maximum of 205 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Standard Fluids | Restricted Fluids
Number analyzed (Participants) | 32 | 32
hours | 45 [26 to 85] | 42 [26 to 69]

2. Secondary Outcome: Duration of ICU Admission
Time Frame: every day until discharge, an average of approximately 8 days and a maximum of 12 days
Measure: Mean (Inter-Quartile Range); unit: calendar days
Arm/Group | Standard Fluids | Restricted Fluids
Number analyzed (Participants) | 32 | 32
calendar days | 8 [5 to 12] | 7 [4 to 10]

3. Secondary Outcome: Time to First Enteral Feed
Time Frame: hour until first enteral feed achieved, an average of approximately 40 hours and a maximum of 100 hours
Measure: Mean (Inter-Quartile Range); unit: hours
Arm/Group | Standard Fluids | Restricted Fluids
Number analyzed (Participants) | 32 | 32
hours | 31 [21 to 51] | 35 [23 to 44]

ADVERSE EVENTS:
Time Frame: Study safety was assessed daily for all enrolled patients. Predetermined indicators of dehydration including daily weight, daily urine output, and daily serum sodium, blood urea nitrogen (BUN), creatinine, glucose, and bilirubin level were monitored.
Description: No patient enrolled in the study experienced an adverse event or unsafe fluid or glycemic balance due to the study protocol.
Arm/Group | Standard Fluids | Restricted Fluids
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

LIMITATIONS AND CAVEATS:
As a small, single center study, our results may not be fully generalizable to the TTN patient population in all hospital types on a national level.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes